CLINICAL TRIAL: NCT03358693
Title: Systematic Profiling of Anti-cytokine Signatures in the Treatment of Chronic Inflammatory Skin Disorders
Brief Title: Molecular Signatures in Inflammatory Skin Disease
Acronym: MSID
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Stephan Weidinger (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Stephan Weidinger, Head, Inflammatory Skin Disease Center, University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Other Study IDs: A100/12; A100/12_A (Other: Ethics Committee Medical Faculty Kiel, Amendment 11MAR2017)
Record Dates: First submitted 2017-11-04; First posted 2017-11-30 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis | interventions — dupilumab; baricitinib; abrocitinib; upadacitinib; tralokinumab; lebrikizumab; nemolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, swabs, tape strips, skin biopsies (only adults)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (13):
- Psoriasis patients receiving Tumor Necrosis Factor (TNF) Inhibitors: Pso_Tumor Necrosis Factor (TNF) Inhibitors
  Interventions: Drug: Anti-TNF
- Psoriasis patients receiving Interleukin (IL)-12/23 Inhibitors: Interleukin (IL)-12/23 Inhibitors
  Interventions: Drug: Anti-IL12/23
- Psoriasis patients receiving Interleukin (IL)-17 Inhibitors: Pso_Interleukin (IL)-17 Inhibitors
  Interventions: Drug: Anti-IL17
- Atopic dermatitis patients receiving dupilumab: Dupilumab
  Interventions: Drug: Dupilumab
- Atopic dermatitis patients receiving lebrikizumab: Brodalumab
  Interventions: Drug: Lebrikizumab
- Atopic dermatitis patients receiving tralokinumab: Tralokinumab
  Interventions: Drug: Tralokinumab
- Atopic dermatitis patients receiving baricitinib: Baricitinib
  Interventions: Drug: Baricitinib
- Atopic dermatitis patients receiving abrocitinib: Abrocitinib
  Interventions: Drug: Abrocitinib
- Atopic dermatitis patients receiving upadacitinib: Upadacitinib
  Interventions: Drug: Upadacitinib
- Psoriasis patients receiving Interleukin (IL)-23 Inhibitors: Interleukin (IL)-23 Inhibitors
  Interventions: Drug: Anti-IL23
- Atopic dermatitis patients receiving Interleukin (IL)-31 Inhibitors: Interleukin (IL)-31 Inhibitors
  Interventions: Drug: Nemolizumab
- Hidradenitis patients receiving Interleukin (IL)-17 Inhibitors: HS_Interleukin (IL)-17 Inhibitors
  Interventions: Drug: Anti-IL17
- Hidradenitis patients receiving Tumor Necrosis Factor (TNF) Inhibitors: HS_Tumor Necrosis Factor (TNF) Inhibitors
  Interventions: Drug: Anti-TNF

INTERVENTIONS:
Drug: Anti-TNF — Subject receives anti-TNF antibodies open-label as per guidelines
  Groups: Hidradenitis patients receiving Tumor Necrosis Factor (TNF) Inhibitors; Psoriasis patients receiving Tumor Necrosis Factor (TNF) Inhibitors
Drug: Anti-IL12/23 — Subject receives anti-IL12/23 antibodies open-label as per guidelines
  Groups: Psoriasis patients receiving Interleukin (IL)-12/23 Inhibitors
Drug: Anti-IL17 — Subject receives anti-IL17 antibodies open-label as per guidelines
  Groups: Hidradenitis patients receiving Interleukin (IL)-17 Inhibitors; Psoriasis patients receiving Interleukin (IL)-17 Inhibitors
Drug: Dupilumab — Subject receives Dupilumab open-label as per guidelines
  Groups: Atopic dermatitis patients receiving dupilumab
Drug: Anti-IL23 — Subject receives anti-IL23 antibodies open-label as per guidelines
  Groups: Psoriasis patients receiving Interleukin (IL)-23 Inhibitors
Drug: Baricitinib — Subject receives Baricitinib open-label as per guidelines
  Groups: Atopic dermatitis patients receiving baricitinib
Drug: Abrocitinib — Subject receives Abrocitinib open-label as per guidelines
  Groups: Atopic dermatitis patients receiving abrocitinib
Drug: Upadacitinib — Subject receives Upadacitinib open-label as per guidelines
  Groups: Atopic dermatitis patients receiving upadacitinib
Drug: Tralokinumab — Subject receives Tralokinumab open-label as per guidelines
  Groups: Atopic dermatitis patients receiving tralokinumab
Drug: Lebrikizumab — Subject receives Lebrikizumab open-label as per guidelines
  Groups: Atopic dermatitis patients receiving lebrikizumab
Drug: Nemolizumab — Subject receives Nemolizumab open-label as per guidelines
  Groups: Atopic dermatitis patients receiving Interleukin (IL)-31 Inhibitors

SUMMARY:
This pilot project intends to examine the utility of a systems medicine approach to identify regulatory networks and their perturbation in psoriasis and atopic dermatitis, and to obtain a comprehensive perspective on disease and disease control by integrating and modelling data across multiple cellular levels and time following specific blockade of single pathophysiological factors through use of licensed biologics during routine care as systems biology challenge. To this end, ultra-deep phenotyping and prospective molecular characterization in short time-intervals and different disease equilibrium states will be carried out in targeted small sets of patients. The different layers and types of clinical and molecular information will then be integrated (integrative personal omics profiling iPOP) for generating insights into disease pathways and for extraction of molecular signatures that correspond to clinical severity scores. It will provide a good starting point for planning future trials aimed at identifying biological patterns useful for guiding targeted treatment.

DETAILED DESCRIPTION:
This is an exploratory study with the aim to identify molecular profiles and signatures in skin and blood that correlate with inflammatory skin disease, disease activity and disease progression, and that are associated with possible disease subtypes/endotypes. Primary target variables are differentially expressed genes (alone or in combination), secondary target variables are genetic, immunological and microbiological signatures. Influencing variables of interest include age of manifestation, disease duration, disease activity/severity, disease progression, comorbidities and therapy/treatment. Obtained biomaterial will be used for molecular profiling including DNA/RNA sequencing, ELISA, mass spectrometry, flow cytometry to identify markers and/or signatures that can correlate with individual disease courses.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with the protocol
* Dermatologist-diagnosed chronic inflammatory skin disease
* Subject receives systemic therapy within routine care (in-label use of biologics)

Exclusion Criteria:

* Subject is unable to provide written informed consent or comply with the protocol.
* Having used immunosuppressive/immunomodulating therapy or phototherapy within 4 weeks before the baseline visit.
* Treatment of selected skin areas to be examined with topical corticosteroid or topical calcineurin inhibitor within 1 week before the baseline visit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic inflammatory skin disease who receive systemic therapy from their treating dermatologist during routine care
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of molecular profiles over time | Baseline and week 2, week 4, week 12, week 52
  Changes of immune cell composition, transcriptome, proteome and microbiome signatures
Changes of molecular profiles associated with disease severity/remission | Baseline and week 2, week 4, week 12, week 52
  Changes of immune cell composition, transcriptome, proteome and microbiome signatures
Changes of molecular profiles associated with treatment | Baseline and week 2, week 4, week 12, week 52
  Changes of immune cell composition, transcriptome, proteome and microbiome signatures
Changes of molecular profiles associated with treatment response | Baseline and week 2, week 4, week 12, week 52
  Changes of immune cell composition, transcriptome, proteome and microbiome signatures

SECONDARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) score | Baseline and week 1, week 2, week 12, week 52
  Clinical severity score
Change in Score of Atopic Dermatitis (SCORAD) | Baseline and week 1, week 2, week 12, week 52
  Clinical severity score
Change in Psoriasis Area and Severity Index (PASI) | Baseline and week 1, week 2, week 12, week 52
  Clinical severity score
Change in Hidradenitis Suppurativa Severity Score (IHS4) | Baseline and week 1, week 2, week 12, week 52
  Clinical severity score

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Weidinger, MD, Principal Investigator — Department of Dermatology, university Hospital Schleswig-Holstein, Campus Kiel
Locations (1):
- Department of Dermatology, University Hospital Schleswig Holstein, Campus Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No